CLINICAL TRIAL: NCT02680184
Title: A Multicenter, Two Part Open-Label, Phase 1B Clinical Study of CMP-001 Administered Either in Combination With Pembrolizumab or as a Monotherapy in Subjects With Advanced Melanoma
Brief Title: Clinical Study of CMP-001 in Combination With Pembrolizumab or as a Monotherapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CMP-001-001
Record Dates: First submitted 2016-01-26; First posted 2016-02-11 (Estimated); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
Keywords: Malignant Melanoma; Stage IV Skin Melanoma; vidutolimod
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Dose-Escalation - CMP-001 and Pembrolizumab (Experimental): Participants will receive up to 5 escalating dose levels (1 milligram [mg], 3 mg, 5 mg, 7.5 mg and 10 mg) of CMP-001 via intratumoral injection according to one of 2 schedules (Schedule A: once weekly for 7 weeks, followed by every 3 weeks thereafter until participant is discontinued; Schedule B: once weekly for 2 weeks, followed by every 3 weeks thereafter until participant is discontinued) in combination with pembrolizumab at its labelled dose and schedule.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab
- Part 1: Dose-Expansion - CMP-001 and Pembrolizumab (Experimental): Participants will receive CMP-001 10 mg via intratumoral injection by Schedule A (once weekly for 7 weeks, followed by every 3 weeks thereafter until participant is discontinued) in combination with pembrolizumab at its labelled dose and schedule. As of 05 October 2018, the dose and schedule for Part 1 Dose Expansion Phase was selected based on all available safety, efficacy and pharmacodynamic data from the Part 1 Dose Escalation Phase. Participants who were enrolled prior to 05 October 2018 to receive CMP-001 doses less than (<) 10 mg will have the option to receive CMP-001 doses up to 10 mg on Schedule A in combination with pembrolizumab.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab
- Part 2: CMP-001 Monotherapy and Crossover to Combination (Experimental): Participants will receive CMP-001 10 mg via intratumoral injection by Schedule A (once weekly for 7 weeks, followed by every 3 weeks thereafter until participant is discontinued). Participants who were enrolled prior to 05 October 2018 to receive CMP-001 doses <10 mg will have the option to receive CMP-001 doses up to 10 mg on Schedule A. Participants with documented progression while on CMP-001 monotherapy treatment will have the option to crossover to the combination treatment of CMP-001 10 mg plus pembrolizumab, at the discretion of the Investigator.
  Interventions: Drug: CMP-001; Drug: Pembrolizumab

INTERVENTIONS:
Drug: CMP-001 — CMP-001 will be administered as per the dose and schedule specified in the respective arms.
  Other Names: vidutolimod
Drug: Pembrolizumab — Pembrolizumab will be administered as per the schedule specified in the respective arms.
  Other Names: Keytruda

SUMMARY:
This study will be conducted in two parts: Part 1 will be conducted using a Dose Escalation and Expansion design. The Part 1 Dose Escalation Phase of this study will identify a safe and tolerable dose to be further evaluated in the Part 1 Dose Expansion phase. Part 2 of the study will be conducted in parallel with the Part 1 Dose Expansion Phase and will evaluate the safety and efficacy of CMP-001 when administered as a monotherapy. A Treatment Extension to assess the safety profile of CMP-001 when given in combination with pembrolizumab or as monotherapy will be available to those who are currently being treated in either Part 1 or Part 2 of this study at the time of protocol Amendment 9, v10.0.

DETAILED DESCRIPTION:
Former Sponsor Checkmate Pharmaceuticals

The primary objective of Part 1 of the study is to determine the recommended Phase 2 dose (RP2D) and schedule of CMP-001 when given in combination with pembrolizumab in participants with advanced melanoma.

The primary objective of Part 2 of the study is to assess and describe the safety profile of CMP-001 when administered as monotherapy.

The primary objective of the Treatment Extension is to assess the safety profile of CMP-001 when given in combination with pembrolizumab or as monotherapy in the Treatment Extension.

Participants enrolled into either Part 1 or Part 2 will continue study treatment as long as they do not experience unacceptable toxicities and when continued treatment, is in the participant's best interest according to the Investigator. Participants may continue therapy beyond progression based upon Investigator judgement of potential benefit.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed diagnosis of metastatic, or unresectable, malignant melanoma. Ocular melanoma participants are not eligible
* Participants who are currently receiving treatment with any anti-programmed cell death-1/programmed death-ligand 1 (anti-PD-1/PD-L1) antibody, either alone or in combination and who are progressing. Participants must have received at least 4 doses of anti-PD-1/PD-L1 before enrolling into the CMP-001-001 study; or
* Participants who have previously received any anti-PD-1/PD-L1 therapy, alone or in combination and progressed, regardless of the best overall response to prior anti-PD-1/PD-L1 based therapy. Participants must have received at least 4 doses of anti-PD-1/PD-L1 (Inclusion criterion for Part 1 only)
* Participants must have at least one tumor lesion with a longest diameter of greater than or equal to (>=)0.5 centimeter (cm) that can be easily palpated or detected by ultrasound to facilitate intratumoral injection of CMP-001 (that is [i.e.], tumor in skin, muscle, subcutaneous tissue or accessible lymph node)
* Participants must have measurable disease by RECIST version 1.1.
* Capable of understanding and complying with protocol requirements
* A life expectancy of greater than 24 weeks at Screening
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Most recent laboratory values (within 3 weeks prior to Week 1 Day 1) before study entry meet the following standards:
* Bone marrow function: neutrophil count >=1,000/cubic millimeter (mm^3); platelet count >=75,000/mm^3 and hemoglobin concentration >8.0 grams per deciliter (g/dL).
* Liver function: total bilirubin less than or equal to (<=) 1.5 times the upper limit of normal (ULN) ranges of each institution, with the following exception: participants with Gilbert Disease serum bilirubin > 3*ULN; and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <=3 times the ULN range of each institution
* Lactate dehydrogenase (LDH) <=2.0 times the ULN range of each institution
* Renal function: serum creatinine <=1.5 times the ULN range of each institution
* The participant must sign a written informed consent form prior to the initiation of any study procedures. Adult participants unable to provide written informed consent on their own behalf will not be eligible for the study

Part 1 Dose Expansion Phase participants must also meet the following inclusion criterion:

• At least one additional lesion that is measurable and is not intended for injection (to allow an assessment of systemic antitumor effect). These lesions not intended for injection may be located in any metastatic site.

Exclusion Criteria:

* Pregnant or breastfeeding
* Received investigational therapy (that is, small molecule or biologic) within 30 days prior to the start of CMP-001 dosing on Week 1 Day 1. Received prior therapy with anti- cytotoxic T-lymphocyte-associated protein 4 (anti-CTLA-4) antibody within 30 days (within 45 days for Part 2 participants) prior to the start of CMP-001 dosing on Week 1 Day 1. However, if an investigational therapy has a short half-life, a reduced wash out period may be acceptable with Sponsor approval
* Known infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). If there is no known or documented history of HIV, Hepatitis B or Hepatitis C, the site is not required to do additional testing for these values at Screening
* Developed autoimmune disorders of Grade 4 while on prior immunotherapy (Exclusion criterion for Part 1 only). Participants who developed autoimmune disorders of Grade <=3 may enroll if the disorder has resolved to Grade <=1 and the participant has been off systemic steroids at doses > 10 milligrams per day (mg/day) for at least two weeks
* Require systemic pharmacologic doses of corticosteroids greater than the equivalent of 10 mg/day prednisone; replacement doses, topical, ophthalmologic and inhalational steroids are permitted. Participants who have a history of adrenal insufficiency and are receiving greater than 10 mg/day corticosteroid may be eligible but only after Sponsor consultation. Participants who are currently receiving steroids at a dose of <=10 mg/day do not need to discontinue steroids prior to enrollment
* Active (i.e., symptomatic or growing) central nervous system (CNS) metastases. However, participants with active CNS metastases are eligible for the trial if

  * the metastases have been treated by surgery and/or radiotherapy,
  * the participant is off corticosteroids >10 mg/day and is neurologically stable for at least 2 weeks prior to Screening
  * brain imaging (by CT, positron emission tomography [PET], MRI, or per site standards) completed within 3 months of screening (required for all participants)
* Any concurrent uncontrolled illness, including mental illness or substance abuse, which in the opinion of the Investigator, would make the participant unable to cooperate or participate in the trial
* Severe uncontrolled cardiac disease within 6 months of Screening, including but not limited to uncontrolled hypertension; unstable angina; myocardial infarction (MI) or cerebrovascular accident (CVA)
* Requires prohibited treatment (i.e., non-protocol specified anticancer pharmacotherapy, surgery or conventional radiotherapy for treatment of malignant tumor)
* Women of child-bearing potential who are unable or unwilling to use an acceptable method of contraception

Main Criteria for Inclusion: Treatment Extension (CMP-001 alone or in combination with pembrolizumab)

* Actively being treated in either Part 1 or Part 2 of this study.
* Subject has signed an additional written ICF for Protocol Amendment 9 (v10.0) prior to receiving the first dose of CMP-001 and/or pembrolizumab in the Treatment Extension. Adult subjects unable to provide written informed consent on their own behalf will not be eligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 199 (Actual)
Dates: Start 2016-04-12 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Part 1: Dose-Escalation Phase: RP2D of CMP-001 When Given in Combination With Pembrolizumab | 21 days (for Schedule A dosing) and 35 days (for Schedule B dosing)
Part 2 Monotherapy: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | From first dose of CMP-001 (Week 1 Day 1) until 30 days after the last CMP-001 injection (up to approximately 3.5 years)
  TEAEs will be evaluated and assigned a grade using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.

SECONDARY OUTCOMES:
Part 1 Dose Escalation and Dose Expansion: Number of Participants With TEAEs | From first dose of CMP-001 (Week 1 Day 1) until 30 days after the last CMP-001 injection (up to approximately 3.5 years)
  TEAEs will be evaluated and assigned a grade using CTCAE version 5.0
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Oral Temperature | From screening up to end of treatment (EOT) (up to approximately 3.5 years)
  Oral temperature should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Respiratory Rate | From screening up to EOT (up to approximately 3.5 years)
  Respiratory rate should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Systolic and Diastolic Blood Pressure | From screening up to EOT (up to approximately 3.5 years)
  Blood pressure should be measured in supine or seated position, following at least 30 minutes of rest.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Body Weight | From screening up to EOT (up to approximately 3.5 years)
  Physical examination included body weight measurement.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Body Mass Index (BMI) | From screening up to EOT (up to approximately 3.5 years)
  Physical examination included BMI measurement.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Number of Participants With Clinically Significant Abnormalities in 12-Lead Electrocardiogram (ECG) Parameters | From screening up to EOT (up to approximately 3.5 years)
  ECG parameters will include heart rate and PR, QRS, QT, and QT corrected for heart rate (QTc) intervals. QT will be corrected using Fridericia's (QTcF) formula. ECG will be performed after the participant has been resting in supine or semi-supine position for at least 5 minutes.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Number of Participants With Clinically Significant Abnormalities in Clinical Laboratory Parameters | From screening up to EOT (up to approximately 3.5 years)
  Clinical laboratory parameters includes serum chemistry, hematology, and urinalysis.
Part 1 Dose Escalation: Concentration of Chemokine IP-10 | Schedule A: Screening, Day 1 of Weeks 1, 3, 7, and Day 2 of Weeks 3, 7; Schedule B: Screening, Day 1 of Weeks 1, 5, 17, and Day 2 of Weeks 5, 17
Part 1 and Part 2: Objective Response Rate (ORR) (Percentage of Participants With Objective Response) as per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 Using Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI) Scans | Baseline until confirmed disease progression (CR or PR) or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 3.5 years)
  ORR will be calculated as the number of participants with a confirmed complete response (CR) or partial response (PR) divided by the number of participants dosed.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Progression-Free Survival (PFS) as per RECIST Version 1.1 Using CT or MRI Scans | From first dose of CMP-001 until disease progression or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 3.5 years)
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Best Overall Response (BOR) Rate (Percentage of Participants With Best Objective Response of CR or PR) as per RECIST Version 1.1 Using CT or MRI Scans | Baseline until confirmed disease progression (CR or PR) or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 3.5 years)
  BOR will be calculated as the number of participants with best response of CR or PR divided by the number of participants dosed.
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Time to Response (TTR) as per RECIST Version 1.1 Using CT or MRI Scans | From first dose of CMP-001 until disease progression or death, whichever occur first (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 3.5 years)
Part 1 Dose Escalation and Dose Expansion, and Part 2 Monotherapy: Duration of Response (DOR) as per RECIST Version 1.1 Using CT or MRI Scans | From the date of first confirmed CR or PR until the first date of recurrent or progressive disease (assessment at every 12 weeks throughout the study from Week 1 Day 1, up to approximately 3.5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (13):
- United States (13):
  - Banner MD Anderson Cancer Center, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - University of California, Los Angeles, Los Angeles, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Georgetown, Washington D.C., District of Columbia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/